CLINICAL TRIAL: NCT02723084
Title: A Randomized, Open-Label, Active Comparator, Multicenter Study to Evaluate the Efficacy and Safety of ABT-493/ABT-530 in Japanese Adults With Genotype 2 Chronic Hepatitis C Virus Infection (CERTAIN-2)
Brief Title: A Study to Evaluate the Efficacy and Safety of ABT-493/ABT-530 in Japanese Adults With Genotype 2 Chronic Hepatitis C Virus Infection
Acronym: CERTAIN-2
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: AbbVie (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: M15-828
Record Dates: First submitted 2016-03-24; First posted 2016-03-30 (Estimated); Results first posted 2019-02-15 (Actual); Last update posted 2021-07-16 (Actual); Status verified 2021-07

CONDITIONS: Chronic Hepatitis C Virus; Hepatitis C Virus
Keywords: Hepatitis C Virus; Non-cirrhotic; Hepatitis C Genotype 2; Chronic Hepatitis C Virus; Hepatitis C
MeSH Terms: conditions — Hepatitis C, Chronic; Hepatitis C | interventions — glecaprevir and pibrentasvir; glecaprevir; pibrentasvir; Sofosbuvir; Ribavirin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Arm A (Experimental): Co-formulated ABT-493/ABT-530 (300 mg/120 mg) administered once daily (QD) for 8 weeks in HCV genotype (GT) 2 -infected, DAA treatment-naïve participants without cirrhosis.
  Interventions: Drug: ABT-493/ABT-530
- Arm B (Active Comparator): sofosbuvir (400 mg) QD co-administered with weight based ribavirin (RBV) 600-1000 mg divided twice daily (BID) for 12 weeks in HCV GT2 -infected, DAA treatment-naïve participants without cirrhosis.
  Interventions: Drug: sofosbuvir (SOF); Drug: ribavirin (RBV)

INTERVENTIONS:
Drug: ABT-493/ABT-530 — Co-formulated tablet
  Other Names: glecaprevir/pibrentasvir; glecaprevir (ABT-493); pibrentasvir (ABT-530)
  Arms: Arm A
Drug: sofosbuvir (SOF) — Tablet
  Arms: Arm B
Drug: ribavirin (RBV) — Capsule
  Arms: Arm B

SUMMARY:
The purpose of this phase 3 study is to evaluate the efficacy and safety of ABT-493/ABT-530 in comparison to sofosbuvir plus ribavirin for 12 weeks in Hepatitis C Virus (HCV) Genotype 2 (GT2) infected participants.

DETAILED DESCRIPTION:
This was a randomized, open-label, active-control, multicenter study to evaluate efficacy, safety, and pharmacokinetics of ABT-493/ABT-530 in chronic HCV GT2-infected direct-acting antiviral agent (DAA) treatment-naïve Japanese adult participants without cirrhosis. The participants were randomized in a 2:1 ratio to ABT-493/ABT-530 for 8 weeks (Arm A) and sofosbuvir plus ribavirin for 12 weeks (Arm B).

ELIGIBILITY:
Inclusion Criteria:

* Females were postmenopausal for at least 2 years prior to screening; surgically sterile or had a vasectomized partner; or, if of childbearing potential and sexually active with a male partner, were currently using at least 1 effective method of birth control at the time of Screening and agreed to practice 1 effective method of birth control from Screening through 30 days after stopping study drug. Sexually active males were surgically sterile or, if sexually active with a female partner of childbearing potential, agreed to practice 1 effective form of birth control from Screening through 30 days after stopping study drug.
* Screening central laboratory result indicating HCV GT-2 infection without co-infection of any other genotype.
* Participant has positive anti-HCV antibody (Ab) and plasma HCV RNA viral load greater than or equal to 1000 IU/mL at Screening Visit.
* Chronic HCV infection defined as one of the following:

  * Positive for anti-HCV Ab and/or HCV RNA at least 6 months before Screening; or
  * A liver biopsy consistent with chronic HCV infection.
* Participant must be HCV treatment-naïve (i.e., patient has not received a single dose of any approved or investigational DAA) and non-cirrhotic. Prior HCV treatment using IFNs with or without ribavirin is acceptable. Previous HCV Interferon (IFN) based treatment must have been completed greater than or equal to 2 months prior to screening.

Exclusion Criteria:

* Females who were pregnant or planned to become pregnant, or breastfeeding or males whose partner was pregnant or planning to become pregnant during the study.
* Recent (within 6 months prior to study drug administration) history of drug or alcohol abuse that could preclude adherence to the protocol in the opinion of the investigator.
* Positive test result at Screening for hepatitis B surface antigen (HBsAg) or anti human immunodeficiency virus antibody (HIV Ab).
* Requirement for and inability to safely discontinue contraindicated medications or supplements at least 2 weeks or 10 half-lives (whichever is longer) prior to the first dose of any study drug.
* Clinically significant abnormalities, other than HCV-infection, based upon the results of a medical history, physical examination, vital signs, laboratory profile, and a 12-lead electrocardiogram (ECG) that make the participant an unsuitable candidate for this study in the opinion of the investigator, including, but not limited to:

  * Uncontrolled diabetes as defined by a glycated hemoglobin (hemoglobin A1C) level > 8.5% at the Screening Visit.
  * Active or suspected malignancy or history of malignancy (other than basal cell skin cancer or cervical carcinoma in situ) in the past 5 years, or any history of hepatocellular carcinoma (HCC).
  * Uncontrolled cardiac, respiratory, gastrointestinal, hematologic, neurologic, psychiatric, or other medical disease or disorder, which is unrelated to the existing HCV infection.
* Any cause of liver disease other than chronic HCV-infection, including but not limited to the following:

  * Hemochromatosis, alpha-1 antitrypsin deficiency, Wilson's disease, autoimmune hepatitis, alcoholic liver disease, or steatohepatitis considered to be the primary cause of the liver disease rather than concomitant/incidental with HCV infection.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 136 (Actual)
Dates: Start 2016-04-08 (Actual); Primary Completion 2017-01-19 (Actual); Study Completion 2017-03-24 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: AbbVie Inc., MD, Study Director — AbbVie

REFERENCES:
- [Background] Toyoda H, Chayama K, Suzuki F, Sato K, Atarashi T, Watanabe T, Atsukawa M, Naganuma A, Notsumata K, Osaki Y, Nakamuta M, Takaguchi K, Saito S, Kato K, Pugatch D, Burroughs M, Redman R, Alves K, Pilot-Matias TJ, Oberoi RK, Fu B, Kumada H. Efficacy and safety of glecaprevir/pibrentasvir in Japanese patients with chronic genotype 2 hepatitis C virus infection. Hepatology. 2018 Feb;67(2):505-513. doi: 10.1002/hep.29510. Epub 2017 Nov 24. PMID 28865152
- [Derived] Naganuma A, Chayama K, Notsumata K, Gane E, Foster GR, Wyles D, Kwo P, Crown E, Bhagat A, Mensa FJ, Otani T, Larsen L, Burroughs M, Kumada H. Integrated analysis of 8-week glecaprevir/pibrentasvir in Japanese and overseas patients without cirrhosis and with hepatitis C virus genotype 1 or 2 infection. J Gastroenterol. 2019 Aug;54(8):752-761. doi: 10.1007/s00535-019-01569-7. Epub 2019 Mar 13. PMID 30868245
- [Derived] Krishnan P, Schnell G, Tripathi R, Beyer J, Reisch T, Dekhtyar T, Irvin M, Xie W, Fu B, Burroughs M, Redman R, Kumada H, Chayama K, Collins C, Pilot-Matias T. Integrated Resistance Analysis of CERTAIN-1 and CERTAIN-2 Studies in Hepatitis C Virus-Infected Patients Receiving Glecaprevir and Pibrentasvir in Japan. Antimicrob Agents Chemother. 2018 Jan 25;62(2):e02217-17. doi: 10.1128/AAC.02217-17. Print 2018 Feb. PMID 29180522
- See also: Related Info — http://www.rxabbvie.com/

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Intent-to-treat population: all participants who received at least 1 dose of study drug.
Period: Overall Study
Arm/Group | Arm A | Arm B
Started | 90 | 46
Completed | 86 | 45
Not Completed | 4 | 1
Not completed — Withdrawal by Subject | 1 | 1
Not completed — Lost to Follow-up | 3 | 0

BASELINE CHARACTERISTICS:
Population: All participants who received at least 1 dose of study drug (ITT population).
Groups:
- Total: Total of all reporting groups
Arm/Group | Arm A | Arm B | Total
Number analyzed (Participants) | 90 | 46 | 136
Age, Continuous [Mean (Standard Deviation); unit: years] | 57.46 (13.07) | 58.89 (13.64) | 57.94 (13.23)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 48 | 25 | 73
  Male | 42 | 21 | 63
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0
  Not Hispanic or Latino | 90 | 46 | 136
  Unknown or Not Reported | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With Sustained Virologic Response 12 Weeks Post-treatment (SVR12): Non-inferiority of Arm A to Arm B
Description: SVR12 was defined as plasma hepatitis C virus ribonucleic acid (HCV RNA) level less than the lower limit of quantification [<LLOQ]) 12 weeks after the last dose of study drug. The primary efficacy endpoint was non-inferiority of the ABT-493/ABT-530 8-week regimen (Arm A) to the sofosbuvir and ribavirin 12 week regimen (Arm B) in SVR12 using a non-inferiority margin of 10% in the intent-to-treat (ITT) population.
Time Frame: 12 weeks after the last actual dose of study drug
Population: Intent-to-treat (ITT) population: all participants who received at least 1 dose of study drug; participants with missing data after backwards imputation were imputed as nonresponders.
Measure: Number; unit: percentage of participants
Arm/Group | Arm A | Arm B
Number analyzed (Participants) | 90 | 46
percentage of participants | 97.8 | 93.5
Statistical Analysis 1: Comparison: Arm A vs Arm B; Difference in SVR12 rates (Arm A - Arm B); Test type: Non-Inferiority — The percentage of participants achieving SVR12 was calculated for each arm and a 2- sided 95% confidence interval (CI) for the difference in SVR12 rates (Arm A minus Arm B) was calculated using the normal approximation to the binomial distribution to assess non-inferiority in SVR12 rates of arm A to arm B. If the lower bound of the CI for the difference was above the noninferiority margin of -10%, then arm A was considered non-inferior to arm B; Risk Difference (RD) = 4.3, 95% CI 2-sided [-3.5 to 12.1] — 95% CI was calculated using the normal approximation to the binomial distribution

2. Secondary Outcome: Percentage of Participants in Arm A With Sustained Virologic Response 12 Weeks Post-treatment (SVR12)
Description: SVR12 was defined as plasma hepatitis C virus ribonucleic acid (HCV RNA) level less than the lower limit of quantification [<LLOQ]) 12 weeks after the last dose of study drug.
Time Frame: 12 weeks after the last actual dose of study drug
Population: All participants who received at least 1 dose of study drug (ITT population); participants with missing data after backwards imputation were imputed as nonresponders.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Arm A
Number analyzed (Participants) | 90
percentage of participants | 97.8 [94.7 to 100.0]

3. Secondary Outcome: Percentage of Participants With With On-treatment Virologic Failure
Description: On-treatment virologic failure was defined as confirmed increase of > 1 log(subscript)10(subscript) IU/mL above the lowest value post-baseline HCV RNA during treatment, confirmed HCV RNA ≥ 100 IU/mL after HCV RNA < LLOQ during treatment, or HCV RNA ≥ LLOQ at end of treatment with at least 6 weeks of treatment. 95% CI was calculated using the Wilson score method.
Time Frame: Treatment Weeks 1, 2, 4, 8 (end of treatment for arm A), and 12 (end of treatment for arm B) or premature discontinuation from treatment
Population: All participants who received at least 1 dose of study drug (ITT population).
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Arm A | Arm B
Number analyzed (Participants) | 90 | 46
percentage of participants | 0 [0.0 to 4.1] | 0 [0.0 to 7.7]

4. Secondary Outcome: Percentage of Participants With Post-Treatment Relapse
Description: Post-treatment relapse was defined as confirmed HCV RNA ≥ LLOQ between the end of treatment and 12 weeks after the last dose of study drug among participants who completed treatment with HCV RNA levels < LLOQ at the end of treatment, excluding participants who were been shown to be re-infected. 95% CI was calculated using the Wilson score method.
Time Frame: From the end of treatment through 12 weeks after the last dose of study drug
Population: All participants who received at least 1 dose of study drug (ITT population).
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Arm A | Arm B
Number analyzed (Participants) | 89 | 45
percentage of participants | 0 [0.0 to 4.1] | 4.4 [1.2 to 14.8]

ADVERSE EVENTS:
Time Frame: Treatment-emergent adverse events (TEAEs) were collected from the time of study drug administration until 30 days after the last dose of study drug (up to 16 weeks). Serious adverse events (SAEs) were collected starting from the time that the informed consent was signed until the end of the study (up to 21 weeks).
Description: TEAEs and Treatment-emergent serious adverse events (TESAEs) are defined as any adverse event (AE) or serious adverse event (SAE) with an onset date that is after the first dose of study drug until 30 days after the last dose of study drug and were collected whether elicited or spontaneously reported by the participant.
Arm/Group | ARM A | ARM B
All-Cause Mortality (participants affected / at risk) | 0/90 | 0/46
Serious Adverse Events (participants affected / at risk) | 2/90 | 2/46
Other Adverse Events (participants affected / at risk) | 20/90 | 26/46
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | ARM A (N=90) | ARM B (N=46)
ANGINA UNSTABLE (Cardiac disorders) | 1 | 0
PNEUMONIA (Infections and infestations) | 0 | 1
CASTLEMAN'S DISEASE (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
PNEUMOTHORAX SPONTANEOUS (Respiratory, thoracic and mediastinal disorders) | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | ARM A (N=90) | ARM B (N=46)
ANAEMIA (Blood and lymphatic system disorders) | 0 | 16
NAUSEA (Gastrointestinal disorders) | 3 | 3
STOMATITIS (Gastrointestinal disorders) | 1 | 3
MALAISE (General disorders) | 5 | 4
NASOPHARYNGITIS (Infections and infestations) | 9 | 5
BLOOD BILIRUBIN INCREASED (Investigations) | 1 | 7
HYPERURICAEMIA (Metabolism and nutrition disorders) | 0 | 3
HEADACHE (Nervous system disorders) | 6 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
AbbVie requests that any investigator or institution that plans on presenting/publishing results disclosure, provide written notification of their request 60 days prior to their presentation/publication. AbbVie requests that no presentation/publication will be instituted until 12 months after a study is completed, or after the first presentation/publication whichever occurs first. A delay may be proposed of a presentation/publication if AbbVie needs to secure patent or proprietary protection.

DOCUMENTS (2):
  • Study Protocol (2016-06-17): https://cdn.clinicaltrials.gov/large-docs/84/NCT02723084/Prot_001.pdf
  • Statistical Analysis Plan (2016-10-31): https://cdn.clinicaltrials.gov/large-docs/84/NCT02723084/SAP_000.pdf